CLINICAL TRIAL: NCT02239601
Title: Chemotherapy - Induced Peripheral Neuropathy (CIPN). Could There be a Role for Physical Therapy Treatment?
Brief Title: Chemotherapy Induced Peripheral Neuropathy. Could Physical Therapy Help Treat Symptoms?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CancerCare Manitoba (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Marshall Pitz, Medical Oncologist and Associate Professor , University of Manitoba, CancerCare Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2014:281
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Peripheral Neuropathy, Secondary to Drugs or Chemicals
Keywords: Physical Therapy; Physiotherapy; Breast Cancer; Chemotherapy Induced Peripheral Neuropathy (CIPN); Nerve gliding exercises; Nerve Entrapment
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases; Nerve Compression Syndromes | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Therapy (Experimental): 4 Physical therapy treatment sessions provided prior to chemotherapy and a home program to continue throughout the trial.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy assessment and treatment for any positive signs of nerve entrapment prior to chemotherapy including nerve gliding exercises, education and splinting. A home program was provided and continued throughout chemotherapy treatment
  Other Names: physiotherapy

SUMMARY:
The cause of Chemotherapy-Induced Peripheral Neuropathy (CIPN) is still unknown. An estimated 55-60% of patients will experience lasting symptoms affecting function for years post-treatment. Physical therapy is an established, effective treatment for entrapped nerves and neuropathic pain. This study sought to identify additional risk factors and provide evidence for the role of physical therapy in the treatment of CIPN.

DETAILED DESCRIPTION:
A common side effect is chemotherapy induced peripheral neuropathy (CIPN). CIPN is a small fibre sensory neuropathy that develops in the hands/feet and worsens with increasing dose and duration of treatment. It impacts the Aβ, Aδ, and C-Fiber function involved in light touch and vibration sense, thermal detection and thermal pain. This results in a variety of positive and/or negative sensory symptoms including hypoesthesia, dysesthesias, hyperalgesia, allodynia and neuropathic pain. Quantitative sensory testing (QST) are a variety of non-invasive tests aimed at quantifying sensory perceptions used in research to clinically assess neuropathy. It is used for sensory detection and pain thresholds for both mechanical and thermal stimuli. QST provides information on large myelinated (Aβ), small thinly myelinated (Aδ) and unmyelinated (C-fiber) function or dysfunction. Deep pressure threshold measured by a pressure algometry stimulates intramuscular afferents, and can be used as a measure of central sensitization when used at a distant site from the site of pain. Aδ fibres transmit cool detection threshold, while warm detection threshold is transmitted by C-fibers. Both noxious heat and noxious cold transmit via C-fiber and Aδ fibers. An increased sensitivity to thermal pain thresholds, results in thermal hyperalgesia.

Physical therapy treatment for nerve disorders is well established in orthopedics and plastic surgery for entrapment neuropathies, neuropathic pain, post-operative nerve repair and regeneration. Nerve gliding exercises are frequently used exercises in physical therapy to improve neural excursion across joints, improve pain and decrease inflammation. Patient reported symptoms (patient questionnaires NPRS, S-LANSS and DASH) and quantitative sensory testing (QST) specifically pain pressure thresholds and vibration were used for the primary purpose in evaluating the role for an upper extremity nerve mobilization physical therapy home program during chemotherapy for the prevention and management of CIPN.

Primary Outcome Measures was the NPRS and reported as those having no vs no pain. Grip strength, Vibration, DASH and S-LANSS were identified outcome measures prior to the trial that would best describe sensory impairment and function for the physical therapy question

Additional QST measures collected included warm/cool, Hot/Cold Pain thresholds that were used with the vibration data to compare quantitative data on the right and left side to evaluate possible a possible dual nerve disorder when combined with surgery as well as identifying different sensory profiles of QST data between those reporting neuropathic pain and non-neuropathic pain using the S-LANSS

A sub analysis of data was completed dividing participants that remained active throughout compared to less active participants to evaluate the effect of exercise on sensory preservation. This was not an intended analysis at the beginning of the trial and these participants were not randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage I-III breast cancer undergoing regular docetaxel treatment either docetaxel-cyclophosphamide (TC) or 5FU-epirubicin-cyclophosphamide-docetaxel (FEC-D).
* Patients that have not had chemotherapy in the past and do not have identified risk factors (listed below in the exclusion criteria).
* All patients must be able to communicate in english or be able to have a translator present at all appointments.

Exclusion Criteria:

* Patients diagnosed with stage IV breast cancer or who have co-morbid conditions that are known to cause peripheral neuropathic symptoms, including previous chemotherapy, exposure to toxins (such as lead), Diabetes, Shingles, B12 deficiency, Alcoholism, Lyme disease, Syphilis, HIV, Hereditary disorders such as Charcot-Marie Tooth.
* Patients not planned to receive Docetaxel therapy.
* Patients who cannot communicate in English and unable to bring an interpreter will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Shay, PhD, Study Director — University of Manitoba; Elizabeth R Hammond, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Rehabilitation Hospital, Health Sciences Centre, 800 Sherbrook St, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen Hammond E, Pitz M, Steinfeld K, Lambert P, Shay B. An Exploratory Randomized Trial of Physical Therapy for the Treatment of Chemotherapy-Induced Peripheral Neuropathy. Neurorehabil Neural Repair. 2020 Mar;34(3):235-246. doi: 10.1177/1545968319899918. Epub 2020 Jan 24. PMID 31976819

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Therapy: 4 Physical therapy treatment sessions provided prior to chemotherapy and a home program to continue throughout the trial.
  Physical Therapy: Physical therapy assessment and treatment for any positive signs of nerve entrapment prior to chemotherapy including nerve gliding exercises, education and splinting. A home program will be provided to continue throughout chemotherapy treatment
- Control: treatment as usual
Period: Overall Study
Arm/Group | Physical Therapy | Control
Started | 29 | 32
Completed | 22 | 26
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control: treatment per usual
- Total: Total of all reporting groups
Arm/Group | Physical Therapy | Control | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 'Pain' or 'no Pain' as Measured by the Numeric Pain Rating Scale
Description: Numeric Pain Rating Scale - pain rating scale 0-10 (0= no pain to 10= most pain imaginable). Reported as percentages of participants with pain (1-10) vs no pain (0)
Time Frame: Regression models of pain reported over time (mid-docetaxel chemotherapy- 6 months post-chemotherapy). Mid-chemotherapy time frame participants were re-assessed after the 2 round of TC and 4th round of FECD.
Measure: Number; unit: percentage of participants
Groups:
- Control: chemotherapy as usual without physical therapy
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 22 | 26
percentage of participants
  Percentage of Participants with Pain (1-10) | 30 | 49
  Percentage of Participants with no pain (0) | 70 | 51
Statistical Analysis 1: Comparison: Physical Therapy vs Control; Test type: Other; p = 0.053, Mixed Models Analysis; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.17 to 1.01]

2. Primary Outcome: Disability of the Arm, Shoulder and Hand (DASH)
Description: A 30 item participant reported questionnaire commonly used to gauge upper limb function. Each item is scored 1-5 with 1 being 'no difficulty' and 5 being 'unable'. Overall score calculated as: [average response (sum of responses divided by number of responses) -1] x 25 to give a score out of 100. Minimum score is 30 with a maximum score of 150. The DASH was chosen because of high test-retest reliability and the responsiveness and construct validity in patients with breast cancer over other quality of life measures. A minimal clinical important difference is a change score of 15. Higher score indicates more impairment to the upper limb
Time Frame: administered on each re-assessment (pre-chemotherapy, mid-way through docetaxel chemotherapy, end of chemotherapy, 6 months post-chemotherapy) and mixed models accounted for all time points
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Physical Therapy: 4 Physical therapy treatment sessions provided prior to chemotherapy along with a home program to continue throughout the trial.
  Physical Therapy: Physical therapy assessment and treatment for any positive signs of nerve entrapment prior to chemotherapy (baseline) including nerve gliding exercises, education and splinting. A home program was provided and continued throughout chemotherapy treatment.
- Control Group: Chemotherapy as usual- no physical therapy intervention
Arm/Group | Physical Therapy | Control Group
Number analyzed (Participants) | 22 | 26
units on a scale | 34 [31 to 45] | 42 [33 to 52]

3. Primary Outcome: Percentage of Participants With Neuropathic Pain Defined by the Self Report Version of Leeds Assessment for Neuropathic Symptoms and Signs (S-LANSS).
Description: a 7 item patient reported questionnaire and was used to confirm the presence of neuropathic pain. The score ranges from 0-19 (no symptoms=0, sever symptoms=19) with a score above 12 indicative of neuropathic pain/symptoms. S-LANSS was chosen because of its' specificity and accuracy in a cancer population. Participants were requested to answer specifically for the hands, not feet.
Time Frame: administered on each re-assessment (Visit 1 - pre-chemotherapy, Visit 2 - half-way through chemotherapy, Visit 3 - end of chemotherapy, Visit 4 - 3 months post-chemotherapy) and mixed models accounted for all time points
Measure: Number; unit: percentage of patients
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 22 | 26
percentage of patients
  Percentage of patients with non-neuropathic visits | 83.9 | 74
  Percentage of Patients with Neuropathic visits | 16.1 | 26

4. Secondary Outcome: Vibration Sensory Analysis
Description: Vibration analysis testing for perception thresholds are specific to Aβ nerve fibres. The TSAII Vibration Sensory Analyzer (VSA): Medoc, Israel, was used. The pulp of the index finger lightly touches the sensor that delivers random and varying vibration amplitudes (µm). The participant responds "yes/no" to sensing the vibration. Vibration perception was selected for its sensitivity and has been suggested to be the first clinical sign of CIPN symptoms and was tested bilaterally. Low score indicates better perception while a higher score is poorer sensation. Perception score reported in micrometers (up to 4cm)
Time Frame: administered on each re-assessment (Visit 1 - pre-chemotherapy, Visit 2 - half-way through chemotherapy, Visit 3 - end of chemotherapy, Visit 4 - 6 months post-chemotherapy) and mixed models accounted for all time points
Measure: Median (Inter-Quartile Range); unit: micrometers (µm)
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 22 | 26
micrometers (µm)
  Left Hand | 0.23 [0.14 to 0.41] | 0.14 [0.04 to 0.31]
  Right Hand | 0.23 [0.14 to 0.41] | 0.23 [0.14 to 0.41]

5. Secondary Outcome: Pain Pressure Thresholds
Description: Pressure Algometry (Somedic AB, Sweden) measured pressure/pain thresholds. A hand-held device applied perpendicular to the muscles being tested. Increasing pressure is applied until the participant determines that the sensation has changed from a feeling of pressure to a feeling of pain and force (Kpa) is recorded. When tested at a distant site from the source of pain this test measures central sensitization. Lower pressure values (more sensitive to noxious stimuli) suggest impaired central pain and/or diminished descending inhibition pathway. The left quadriceps muscle was tested as a measure of central sensitization.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: kpa
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 22 | 26
kpa | 923 (383) | 744 (285)

6. Secondary Outcome: Grip Strength
Description: Hand Dynamometry records grip strength in kgs and was used as a measure of function (3 trials). The dominant hand was tested using the Jamar dynamometer (Patterson medical, USA) in the 2nd handle position. All 48 participants were right handed.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: kgs
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 22 | 26
kgs | 27.2 (5.53) | 21.8 (4.26)

7. Post Hoc Outcome: Vibration Sensory Outcome Stratified by Patient Activity Level
Description: Measuring Activity Participants were asked about their level of exercise per week at each assessment visit. Participants were considered active if they reported engaging in any form of moderate activity at least 4 times a week (consistent with recommended physical activity guidelines beyond activities of daily living such as walking to the bus or walking the dog around the block) at least 4 times per week on at least 3 out of 4 reassessment visits. Types of reported activities included cycling, running, yoga, swimming, Zumba, dance classes, and tennis. Walking was included if it was at least 30 minutes at a moderate pace. This sub-analysis re-defined the groups as 'active' and 'less active' for the comparison of vibration QST data. This was done to observe the possible impact of exercise on sensory preservation
Time Frame: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: micrometers (µm)
Groups:
- Active: Patients that reported being active a least 4 days per week (30 minutes minimum) on 2 or more of the 4 re-assessment visits
- Less Active: Any exercise that falls below the cut-off for active
Arm/Group | Active | Less Active
Number analyzed (Participants) | 15 | 33
micrometers (µm)
  Vibration Left Hand | 0.08 [0.04 to 0.14] | 0.23 [0.13 to 0.42]
  Vibration Right Hand | 0.14 [0.04 to 0.23] | 0.24 [0.14 to 0.49]

ADVERSE EVENTS:
Time Frame: Each participant was followed from one week prior to initiation of chemotherapy to 6 months post-chemotherapy. Because of delays, alterations of schedules, patients were followed on average between 8-12 months. Re-assessment data was collected 2 weeks after mid and post chemotherapy visits and the 3 and 6 month visits where scheduled from their last chemotherapy. This is slightly different for each participant due to delays, hospital admissions, etc....
Description: Accrual has stopped and all treatment and follow-up has been completed and the study is closed.
Arm/Group | Physical Therapy | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT02239601/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02239601/Prot_SAP_001.pdf